CLINICAL TRIAL: NCT02834377
Title: Individualized Goal-directed Hemodynamic Therapy Targeting Preoperatively Assessed Personal Cardiac Output Values in Patients Undergoing High-risk Surgical Procedures: a Prospective and Randomized Clinical Trial
Brief Title: Personalized Hemodynamic Therapy in Patients Undergoing High-risk Surgery
Acronym: TAPIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAPIR-1.0
Record Dates: First submitted 2016-06-01; First posted 2016-07-15 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Complications
Keywords: Cardiac Output; Hemodynamics; Perioperative Care
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment algorithm (Experimental): Patients allocated to the study group will be connected to a cardiac output monitor. An initial haemodynamic assessment will be performed at the beginning of surgery and at regular time intervals (every 15 minutes) during surgery. The personal cardiac output value is targeted.
  Interventions: Other: Treatment algorithm targeting individual cardiac output
- Standard of Care (No Intervention): Patients allocated to the control group will receive the standard care of the hospital.

INTERVENTIONS:
Other: Treatment algorithm targeting individual cardiac output
  Arms: Treatment algorithm

SUMMARY:
The purpose of this study is to evaluate the effectiveness of using the personal preoperatively assessed cardiac output in high-risk patients to guide perioperative administration of fluids and vasoactive drugs on predefined postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years undergoing a major abdominal procedure (including general, urological, gynaecological, and vascular) with an expected duration of surgery ≥ 90 min or presumed blood loss exceeding 1,000 mL (e.g., intrabdominal vascular surgery) and ≥ 1 of the following high-risk criteria:
* acute or chronic renal impairment (serum creatinine ≥ 1.3 mg/dL)
* predefined risk factors for cardiac or respiratory complications
* Immunodeficiency due to a therapy (e.g., immunosuppressants, chemotherapy, radiation, long-term or high-dose steroids)
* Immunodeficiency due to specific diseases (e.g., leukaemia, lymphoma, AIDS)
* severe liver impairment (biopsy proven liver cirrhosis plus 1 of the following: portal hypertension or history of upper gastrointestinal bleeding due to portal hypertension or previous episodes of hepatic insufficiency/hepatic encephalopathy/hepatic coma
* Age ≥ 80 years

Exclusion Criteria:

* Age <18 years
* Pregnancy
* surgery for palliative treatment
* emergency procedure
* refusal of consent
* participation in another randomized controlled trial
* failure to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Number of study participants with at least one complication of a composite of 30-day postinterventional complications | up tp 90 days after study enrollment
  composite of 30-day postinterventional complications defined according to the ESA-ESICM guidelines for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine (acute kidney injury stage 1 or higher [KIDGO]; ARDS; anastomotic breakdown [moderate and severe]; arrhythmia [severe]; cardiac arrest; cardiogenic pulmonary oedema [severe]; deep vein thrombosis [moderate and severe]; delirium; GI bleeding [severe]; Infection, source uncertain [severe]; bloodstream infection [severe]; myocardial infarction [severe]; pneumonia [severe]; paralytic ileus [severe]; postoperative haemorrhage [severe]; pulmonary embolism [severe]; stroke [severe]; superficial, deep, organ/space surgical site infection [severe]; urinary tract infection [severe]; death)

SECONDARY OUTCOMES:
7-day-mortality | up to 7 days after study enrollment
30-day-mortality | up to 30 days after study enrollment
90-day-mortality | up to 90 days after study enrollment
ICU length of stay | up to 90 days after study enrollment
hospital length of stay | up to 90 days after study enrollment
postoperative morbidity survey on days 3, 7, 14, 30 | up to 90 days after study enrollment
postoperative cognitive dysfunction | up to 90 days after study enrollment
  from day 3 after surgical intervention
Biomarkers of the vascular function as prognostic parameters for immunological complications (syndecan 1, sphingosine 1-phosphate, asymmetric dimethylarginine [ADMA], symmetric dimethylarginine [SDMA], arginine, homoarginine | up to 90 days after study enrollment
perioperative changes of primary metabolites [e. g. citric acid cycle, glycolysis, amino acids metabolism], lipid and phospholipid mediators | up to 90 days after study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Saugel, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf; Julia Wagner, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Klinik und Poliklinik für Anästhesiologie, Zentrum für Anästhesiologie und Intensivmedizin, Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicklas JY, Diener O, Leistenschneider M, Sellhorn C, Schon G, Winkler M, Daum G, Schwedhelm E, Schroder J, Fisch M, Schmalfeldt B, Izbicki JR, Bauer M, Coldewey SM, Reuter DA, Saugel B. Personalised haemodynamic management targeting baseline cardiac index in high-risk patients undergoing major abdominal surgery: a randomised single-centre clinical trial. Br J Anaesth. 2020 Aug;125(2):122-132. doi: 10.1016/j.bja.2020.04.094. PMID 32711724